CLINICAL TRIAL: NCT04279457
Title: Single-Center Prospective Study to Investigate the Difference in the Incidence of Contrast-Induced Nephropathy in High-Risk Patients With the Use of the Dye-Vert Plus System
Acronym: Dye-Vert Plus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Aravinda Nanjundappa, Professor, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-637
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: AKI (Acute Kidney Injury) Due to Trauma
MeSH Terms: conditions — Acute Kidney Injury | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Design:
  This is a prospective randomized controlled trial.
Masking Description: The investigators will randomize into each arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standardized Hydration protocol (Active Comparator): These cases will follow Charleston Area Medical Centers standard Hydration protocol
  Interventions: Other: Standardized hydration protocol
- Hydration + Device (Active Comparator): These cases will follow Charleston Area Medical Centers standard hydration protocol plus use the DyeVert Plus System
  Interventions: Device: DyeVert Plus System

INTERVENTIONS:
Device: DyeVert Plus System — The DyeVert Plus System also contains a reusable Contrast Monitoring Wireless Display (CMW) which communicates with the Dye-Vert Plus Disposable to allow real-time monitoring and display of contrast volumes manually injected compared to a predefined, physician-entered contrast usage threshold throughout the procedure. At the end of the procedure, the CMW displays total procedure contrast volume used (mL), % of physician specified limit , total procedure contrast volume saved (mL), and % contrast saved
  Arms: Hydration + Device
Other: Standardized hydration protocol — hydration protocol based up on the Poseidon protocol
  Arms: Standardized Hydration protocol

SUMMARY:
Coronary angiography (CAG) for diagnostic or therapeutic purposes such as percutaneous coronary intervention (PCI) is one of the common procedures which require the use of intravenous contrast media. The reported incidence of contrast induced nephropathy (CIN) in high-risk patients following CAG varies from 10% to 30%. The high rate of CIN in post-PCI patients could be related either to the patient (advanced age, previous CKD, diabetes, dehydration, and concomitant use of other nephrotoxic drugs) or procedure related (intra-arterial route of administration, use of high osmolar contrast media, repeated exposure to contrast within 48 hours, volume of contrast used). Several strategies to prevent or treat CIN have been developed, including hydration, N-acetyl-cysteine, statins, ascorbic acid, bicarbonate, aminophylline, forced diuresis, renal replacement therapy, and choice of low-osmolarity or alternative agents, but one of the most obvious means is to minimize contrast volume. The DyeVert plus Contrast Reduction System, is designed to lower the amount of contrast dye the kidneys are exposed to during a procedure. Because the amount of contrast dye is precisely controlled. The purpose of this prospective study is to understand how the monitoring system of Dye-Vert Plus will impact Acute Kidney Injuries rates in high-risk patients undergoing cardiac catheterization when used in conjunction with a standardized hydration policy.

DETAILED DESCRIPTION:
Coronary angiography (CAG) for diagnostic or therapeutic purposes such as percutaneous coronary intervention (PCI) is one of the common procedures associated with Contrast-induced nephropathy (CIN). The reported incidence of contrast induced nephropathy (CIN) in high-risk patients following CAG varies from 10% to 30%1. The development of CIN after diagnostic coronary angiography and/or percutaneous coronary intervention (PCI) is associated with prolonged hospitalization and a remarkable increase in morbidity, early and late mortality and costs. The high rate of CIN in post-PCI patients could be related either to the patient (advanced age, previous CKD, diabetes, dehydration, and concomitant use of other nephrotoxic drugs) or procedure related (intra-arterial route of administration, use of high osmolar CM, repeated exposure to contrast within 48 h, volume of contrast used, etc.)2-5. Several strategies to prevent or treat CIN have been developed, including hydration, N-acetyl-cysteine, statins, ascorbic acid, bicarbonate, aminophylline, forced diuresis, renal replacement therapy, and choice of lowosmolarity or alternative agents, but one of the most obvious means is to minimize contrast volume. Patients that have a serum creatinine of > 1.5mg/dl and an eGFR < 60ml/min might be at higher risk for AKIs. In quarter one of 2018, CAMC's in-hospital risk-adjusted acute kidney injury for patients undergoing PCI was 10.64, and the US 50th percentile was 6.476. The goal of this study is to reduce in-hospital risk-adjusted acute kidney injury for patients undergoing PCI, below the US 50th, percentile-based NCDR quarterly results of the Cath-PCI registry by quarter one of 2020.

CIN is one of the leading causes of acute kidney injury at Charleston Area Medical Center it is imperative to take steps to prevent it. CIN is associated with a 13% increase in one- year mortality rate when comparing patients without CIN. Studies have also shown an increase in inpatient length of stay and substantial increase cost for patients who experienced CIN. The economic burden associated with CIN is high, the average in-hospital cost of CIN is $10,345 7. Adopting targeted interventions will reduce the incidence of CIN and the overall economic burden at Charleston Area Medical Center.

This trial is aimed at observing whether the use of the monitoring system Dye-Vert PLUS in conjugation with implementing a pre-hydration protocol on patients with high risk for CIN admitted for cardiac angiography and/or interventional cath lab procedures may reduce the incidence of CIN. An additional aim of the study will be to assess if use of the Dye-Vert PLUS monitoring system reduces the use of mean contrast media given in high-risk patients. Additional aims of this initiative will be to evaluate contrast-related complications, such as hypersensitivity reactions, as well as the associated impact of contrast-related complications on hospital health 3 care economics. This initiative will strive to incorporate clinical practice guidelines from SCAI Expert Consensus Statement: 2016 Best Practices in the Cardiac Catheterization Laboratory related to patient risk screening, pre-procedure hydration, and minimizing contrast media dose used.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. 18 years of age or older
  2. Scheduled to undergo CAG and/or PCI
  3. Baseline estimated glomerular filtration rate (eGFR) of ≥20 and ≤60 mL/ min/1.73 m2
  4. Serum creatinine > 1.5mg/dl
  5. Obtaining a Cardiac catheterization.
  6. HTN/Diabetes
  7. Inpatient and outpatient

Exclusion Criteria:

* Exclusion criteria:

  1. 91 years of age or older
  2. Serum creatinine < 1.5mg/dl
  3. eGFR > 60ml/min
  4. Pregnancy
  5. Dialysis
  6. Dye Allergy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1802 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-03 (Estimated)

PRIMARY OUTCOMES:
Monitoring of AKI | 3 days
  Determined by GFR levels

CONTACTS AND LOCATIONS:
Locations (1):
- CAMC Health Education and Research Institute, Charleston, West Virginia, United States